CLINICAL TRIAL: NCT06219486
Title: Use of D-dimers in the Emergency Department to Identify Adult Patients at Very Low Risk of Mortality for Fast-track Treatment - a Randomized Controlled Study
Brief Title: The Safe Fast Track Study
Acronym: SafeFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Slagelse Sygehus (Other); Holbaek Sygehus (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: The SafeFT-study
Record Dates: First submitted 2023-12-10; First posted 2024-01-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Emergency Department; Non-specific Complaints
Keywords: D-dimer; Fast track; emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Usual care
- Intervention (Experimental): Use of D-dimer to guide care of the patient
  Interventions: Diagnostic Test: D-dimer

INTERVENTIONS:
Diagnostic Test: D-dimer — The investigators will measure a D-dimer test on participants and randomize on informing the physician on the value.
  Arms: Intervention

SUMMARY:
Emergency departments (ED) internationally are treating an increasing number of patients.

Most require hospital services but some could be better cared for on alternative pathways.

D-dimer has some unique properties. It is non-specific and is elevated in many acute condi- tions; but conversely remains normal in the absence of significant disease. Previous studies have shown that having a normal D-dimer on arrival to the emergency department is associated with a very low risk of 30-day all-cause mortality.

The investigators propose a multicenter randomized controlled trial using D-dimer to identify patients at low risk and test if providing this information will change time to discharge disposition by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Able to provide oral and written informed consent in Danish
* Blood tests ordered on arrival as part of standard of care
* Ambulatory on arrival or walking to the ambulance (i.e., stable independent gait)
* Normal vital signs (i.e., National Early Warning Score < 3)

Exclusion Criteria:

* Unstable condition requiring immediate care in the resuscitation area
* Triage level red (i.e., the most urgent patients)
* Trauma (minor and major) patients
* High likelihood of requiring a D-dimer analysis on clinical indications during the current hospital contact (e.g., suspected venous thromboembolic disease) that will be ordered on arrival regardless of this study
* Previous participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1538 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | From arrival to physician decision within 4 hours of arrival
  Length of initial emergency department stay (i.e., time from arrival to the emergency department to decision to discharge home or transfer to another department is made (as reported from the treating physician to the study nurse)).

SECONDARY OUTCOMES:
7- and 30-day all-cause mortality from arrival | From arrival until 30-days later
  7- and 30-day all-cause mortality from arrival
Hospital length of stay | From arrival until final discharge within 1 month
  Hospital length of stay
Re-contacts to the emergency department within 30 days from arrival for any reason | From arrival until 30-days later
  Re-contacts to the emergency department within 30 days from arrival for any reason

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Esbjerg Hospital, Esbjerg, Syd
  - Odense University Hospital, Odense, Syd

IPD SHARING:
Plan to Share IPD: No
Not allowed due to Danish law

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT06219486/SAP_000.pdf